CLINICAL TRIAL: NCT04233879
Title: A Phase 3 Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate the Antiretroviral Activity, Safety, and Tolerability of Doravirine/Islatravir Once-Daily in HIV-1 Infected Treatment-Naïve Participants
Brief Title: Study of Doravirine/Islatravir (DOR/ISL 100 mg/0.75 mg) to Evaluate the Antiretroviral Activity, Safety, and Tolerability in Treatment-Naïve Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Infection (MK-8591A-020)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591A-020; MK-8591A-020 (Other: MSD Protocol Number); jRCT2031210024 (Registry Identifier: jRCT); 2019-000590-23 (EudraCT Number)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine; islatravir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: doravirine/islatravir (DOR/ISL) (Experimental): Treatment-naïve participants living with human immunodeficiency virus-1 (HIV-1) that had not received ≤10 days of prior antiretroviral therapy received blinded fixed dose combination (FDC) Doravirine/Islatravir (DOR/ISL) (100 mg doravirine [DOR]/0.75 mg islatravir [ISL]) and placebo to Bictegravir/Tenofovir Alafenamide/Emtricitabine (BIC/FTC/TAF) once daily (QD) from Day 1 to Week 96, and open-label DOR/ISL up to Week 144. At Week 144, participants who consent to enter the optional open-label study extension continued to receive open-label QD FDC of DOR/ISL (100 mg/0.75 mg) for an additional 24 weeks, up to Week 168.
  Interventions: Drug: DOR/ISL; Drug: Placebo to BIC/FTC/TAF
- Group 2: bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) (Active Comparator): Treatment-naïve participants living with HIV-1 that had not received ≤10 days of prior antiretroviral therapy received blinded BIC/FTC/TAF (50 mg bictegravir [BIC], 200 mg emtricitabine [FTC], 25 mg tenofovir alafenamide [TAF]) and placebo to FDC DOR/ISL QD from Day 1 to Week 96, and open-label BIC/FTC/TAF up to Week 144. At Week 144, participants who consent to enter the optional open-label study extension continued to receive QD BIC/FTC/TAF (50 mg/200 mg/25 mg) for an additional 24 weeks, up to Week 168.
  Interventions: Drug: BIC/FTC/TAF; Drug: Placebo to DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — 100 mg DOR/0.75 mg ISL FDC single tablet taken once daily by mouth.
  Other Names: MK-8591A; Doravirine/islatravir
  Arms: Group 1: doravirine/islatravir (DOR/ISL)
Drug: BIC/FTC/TAF — BIC/FTC/TAF 50/200/25 mg FDC single tablet taken once daily by mouth.
  Other Names: Bictegravir/emtricitabine/tenofovir alafenamide
  Arms: Group 2: bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF)
Drug: Placebo to BIC/FTC/TAF — Placebo single tablet matched to BIC/FTC/TAF taken by mouth.
  Arms: Group 1: doravirine/islatravir (DOR/ISL)
Drug: Placebo to DOR/ISL — Placebo single tablet matched to DOR/ISL taken by mouth.
  Arms: Group 2: bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF)

SUMMARY:
This is a phase 3, randomized, controlled, double-blind, multisite clinical study of a once-daily fixed dose combination (FDC) of 100 mg doravirine/0.75 mg islatravir (DOR/ISL [also known as MK-8591A]) in treatment-naïve participants living with human immunodeficiency virus type-1 (HIV-1) infection. The primary objectives are to evaluate the antiretroviral activity, safety, and tolerability of DOR/ISL compared to bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF). The primary hypothesis is that DOR/ISL is noninferior or superior to BIC/FTC/TAF treatment based on the percentage of participants with HIV-1 ribonucleic acid (RNA) <50 copies/mL at Week 48.

DETAILED DESCRIPTION:
Double-blind treatment with the assigned intervention occurs from Day 1 to Week 96, followed by an open-label portion up to Week 144. Participants who benefit from treatment in the opinion of the Investigator may continue their assigned intervention up to Week 168 (or until they have the option to enroll in a DOR/ISL 100 mg/0.25 mg study, whichever is sooner).

ELIGIBILITY:
Inclusion Criteria:

* Is human immunodeficiency virus type 1 (HIV-1) positive
* Is naïve to antiretroviral therapy (ART) defined as having received ≤10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection including prevention of mother-to-child transmission up to 1 month prior to screening.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) Is not a woman of childbearing potential (WOCBP); 2) Is a WOCBP and using an acceptable contraceptive method, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis); 3) A WOCBP must have a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours before the first dose of study intervention; 4) If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required

Exclusion Criteria:

* Has human immunodeficiency virus type 2 (HIV-2) infection
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has an active diagnosis of hepatitis due to any cause, including active hepatitis B virus (HBV) infection (defined as hepatitis B surface antigen [HBsAg]-positive or hepatitis B virus deoxyribonucleic acid [HBV DNA]-positive)
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma
* Has a history or current evidence of any condition (including active tuberculosis infection), therapy, laboratory abnormality or other circumstance (including drug or alcohol use or dependence) that might, in the opinion of the investigator, confound the results of the study or interfere with the participant's participation for the full duration of the study
* Has been treated for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or any prohibited therapy from 45 days prior to Day 1 through the study intervention period
* Is currently participating in or has participated in a clinical study with an investigational compound or device from 45 days prior to Day 1 through the study intervention period
* Has a documented or known virologic resistance to any approved HIV-1 reverse transcriptase inhibitor, or any study intervention
* Has exclusionary laboratory values within 45 days prior to Day 1
* Is female and is expecting to conceive or donate eggs at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (95):
- United States (17):
  - University of Alabama at Birmingham 1917 Research Clinic ( Site 5610), Birmingham, Alabama
  - Pueblo Family Physicians ( Site 5606), Phoenix, Arizona
  - Ruane Clinical Research Group, Inc. ( Site 5624), Los Angeles, California
  - Midway Immunology and Research ( Site 5622), Ft. Pierce, Florida
  - The Kinder Medical Group ( Site 5615), Miami, Florida
  - Floridian Clinical Research, LLC ( Site 5625), Miami Lakes, Florida
  - Orlando Immunology Center ( Site 5613), Orlando, Florida
  - CAN Community Health ( Site 5627), Sarasota, Florida
  - Triple O Research Institute, P.A. ( Site 5621), West Palm Beach, Florida
  - Columbus Regional Research Institute ( Site 5616), Columbus, Georgia
  - Infectious Disease Specialists Of Atlanta PC ( Site 5608), Decatur, Georgia
  - Hennepin Healthcare-Hennepin Healthcare-ID ( Site 5633), Minneapolis, Minnesota
  - Kansas City CARE Clinic ( Site 5607), Kansas City, Missouri
  - University of Pennsylvania ( Site 5630), Philadelphia, Pennsylvania
  - Saint Hope Foundation, Inc. ( Site 5629), Bellaire, Texas
  - North Texas ID Consultants, PA ( Site 5604), Dallas, Texas
  - Texas Centers for Infectious Disease Associates P.A. ( Site 5619), Fort Worth, Texas
- Argentina (5):
  - Helios Salud S.A. ( Site 5802), Buenos Aires, Buenos Aires F.D.
  - IDEAA Foundation ( Site 5807), Buenos Aires, Buenos Aires F.D.
  - Fundación Huesped ( Site 5801), C.a.b.a, Buenos Aires F.D.
  - Instituto CAICI ( Site 5803), Rosario, Santa Fe Province
  - Instituto Oulton ( Site 5804), Córdoba
- Canada (4):
  - Hamilton Health Sciences- Urgent Care Centre-SIS Clinic ( Site 5703), Hamilton, Ontario
  - Toronto General Hospital - University Health Network ( Site 5705), Toronto, Ontario
  - Clinique Medicale L Actuel ( Site 5714), Montreal, Quebec
  - McGill University Health Center - Research Institute-CVIS Clinical Research Unit ( Site 5702), Montreal, Quebec
- Chile (6):
  - Clinica Universidad Catolica del Maule ( Site 5909), Talca, Maule Region
  - Clinica Arauco Salud ( Site 5900), Santiago, Region M. de Santiago
  - Hospital Clinico de la Universidad Catolica ( Site 5903), Santiago, Region M. de Santiago
  - Fundacion Arriaran ( Site 5901), Santiago, Region M. de Santiago
  - Centro Cardiovascular Cardiosur ( Site 5907), Santiago, Region M. de Santiago
  - Hospital Dr. Hernan Henriquez Aravena ( Site 5905), Temuco, Región de la Araucanía
- Colombia (3):
  - Hospital Universitario San Ignacio ( Site 6005), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 6006), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 6001), Cali, Valle del Cauca Department
- France (10):
  - A.P.H. Paris. Hopital Bichat Claude Bernard ( Site 6124), Paris, Ain
  - Hopital de la Croix-Rousse ( Site 6127), Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Regional du Orleans ( Site 6108), Orléans, Centre-Val de Loire
  - Hopital Francois Mitterrand ( Site 6119), Dijon, Cote-d Or
  - CHU de Bordeaux. Hopital Pellegrin ( Site 6116), Bordeaux, Gironde
  - Centre Hospitalier de Tourcoing ( Site 6100), Tourcoing, Nord
  - Hopital Avicenne ( Site 6102), Bobigny, Seine-Saint-Denis
  - A.P.H. Paris, Hopital Saint Louis ( Site 6114), Paris
  - Hopital Saint-Antoine ( Site 6113), Paris
  - Hopital Pitie Salpetriere ( Site 6111), Paris
- Germany (7):
  - Universitaetsklinik Freiburg ( Site 6206), Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum der LMU München ( Site 6204), Munich, Bavaria
  - MVZ Munchen am Goetheplatz ( Site 6202), Munich, Bavaria
  - Infektiologikum ( Site 6201), Frankfurt am Main, Hesse
  - Universitaetsklinikum Bonn ( Site 6200), Bonn, North Rhine-Westphalia
  - EPIMED- Ges. f. epidemiolog. u. klin. Forschung in der Medizin mbH ( Site 6208), Berlin
  - Universitaetsklinikum Hamburg- Eppendorf (UKE) ( Site 6210), Hamburg
- Israel (5):
  - Rambam Medical Center ( Site 6701), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 6702), Jerusalem
  - Chaim Sheba Medical Center. ( Site 6704), Ramat Gan
  - Kaplan Medical Center ( Site 6700), Rehovot
  - Sourasky Medical Center ( Site 6705), Tel Aviv
- Italy (12):
  - A.O.R.N. dei Colli - Ospedale Cotugno ( Site 6407), Napoli, Campania
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 6404), Modena, Emilia-Romagna
  - ASST Papa Giovanni XXIII ( Site 6411), Bergamo, Lombardy
  - Ospedale San Gerardo ASST Monza ( Site 6412), Monza, Monza E Brianza
  - Ospedale Amedeo di Savoia ( Site 6414), Turin, Piedmont
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico ( Site 6401), Milan
  - Salute San Raffaele ( Site 6402), Milan
  - Azienda Ospedaliera San Paolo ( Site 6403), Milan
  - ASST Fatebenefratelli-Ospedale Sacco ( Site 6400), Milan
  - IRCCS Policlinico San Matteo ( Site 6410), Pavia
  - Azienda USL di Pescara-Presidio Ospedaliero di Pescara ( Site 6413), Pescara
  - Istituto Nazionale per Le Malattie Infettive Lazzaro Spallanzani ( Site 6405), Roma
- Japan (5):
  - National Hospital Organization Nagoya Medical Center ( Site 6903), Nagoya, Aichi-ken
  - Kumamoto University Hospital ( Site 6905), Kumamoto
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research ( Site 69, Osaka
  - Tokyo Medical University Hospital ( Site 6904), Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 6901), Tokyo
- South Africa (8):
  - JOSHA Research ( Site 6605), Bloemfontein, Free State
  - Chris Hani Baragwanath Hospital - ICU ( Site 6608), Johannesburg, Gauteng
  - Wits Health Consortium. Clinical HIV Research Unit ( Site 6614), Johannesburg, Gauteng
  - Ezintsha ( Site 6609), Johannesburg, Gauteng
  - Wentworth Hospital ( Site 6607), Durban, KwaZulu-Natal
  - Family Clinical Research Unit (Fam-Cru)-Adult Infectious Diseases ( Site 6617), Cape Town, Western Cape
  - Desmond Tutu HIV Foundation Clinical Trial Unit ( Site 6613), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 6603), Mbekweni, Paarl, Western Cape
- Spain (10):
  - Hospital General de Elche ( Site 6308), Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol ( Site 6301), Badalona, Barcelona
  - Hospital Universitari de Bellvitge ( Site 6312), LHospitalet de Llobregat, Barcelona
  - Hospital Vall D Hebron ( Site 6302), Barcelona, Catalonia
  - Hospital Clinic i Provincial ( Site 6300), Barcelona, Catalonia
  - Hospital General Universitario Gregorio Maranon ( Site 6303), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 6307), Madrid
  - Hospital Universitario 12 de Octubre ( Site 6305), Madrid
  - Hospital Universitario La Paz ( Site 6304), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 6309), Málaga
- Taiwan (3):
  - Kaohsiung Veterans General Hospital ( Site 7102), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 7101), Tainan
  - National Taiwan University Hospital ( Site 7100), Taipei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Rockstroh JK, Paredes R, Cahn P, Molina JM, Sokhela SM, Hinestrosa F, Kassim S, Cunningham D, Ghosn J, Bogner JR, Gatanaga H, Asante-Appiah E, Zhang Y, Nwoke U, Klopfer SO, Eves K, Squires K, Correll T, Fox MC, Pisculli ML. Doravirine/Islatravir (100/0.75 mg) Once-Daily Compared With Bictegravir/Emtricitabine/Tenofovir Alafenamide as Initial HIV-1 Treatment: 48-Week Results From a Phase 3, Randomized, Controlled, Double-Blind, Noninferiority Trial. Clin Infect Dis. 2025 Sep 16;81(2):322-332. doi: 10.1093/cid/ciaf077. PMID 40079835
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment-naïve participants living with Human Immunodeficiency Virus-1 (HIV-1) that had not received ≤10 days of prior antiretroviral therapy were enrolled.
Pre-assignment Details: A total of 599 participants were randomized in the study and 597 received at least 1 dose of study intervention. The safety analyses were conducted using all participants as treated population, which included all randomized participants who received at least 1 dose of study intervention.
Groups:
- Group 1: DOR/ISL: Treatment-naïve participants living with human immunodeficiency virus-1 (HIV-1) that had not received ≤10 days of prior antiretroviral therapy received blinded fixed dose combination (FDC) Doravirine/Islatravir (DOR/ISL) (100 mg doravirine [DOR]/0.75 mg islatravir [ISL]) and placebo to Bictegravir/Tenofovir Alafenamide/Emtricitabine (BIC/FTC/TAF) once daily (QD) from Day 1 to Week 96, and open-label DOR/ISL up to Week 144. At Week 144, participants who consent to enter the optional open-label study extension continued to receive open-label QD FDC of DOR/ISL (100 mg/0.75 mg) for an additional 24 weeks, up to Week 168.
- Group 2: BIC/FTC/TAF: Treatment-naïve participants living with HIV-1 that had not received ≤10 days of prior antiretroviral therapy received blinded BIC/FTC/TAF (50 mg bictegravir [BIC], 200 mg emtricitabine [FTC], 25 mg tenofovir alafenamide [TAF]) and placebo to FDC DOR/ISL QD from Day 1 to Week 96, and open-label BIC/FTC/TAF up to Week 144. At Week 144, participants who consent to enter the optional open-label study extension continued to receive QD BIC/FTC/TAF (50 mg/200 mg/25 mg) for an additional 24 weeks, up to Week 168.
Period: Base Study (Day 1 to Week 144)
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Started | 298 | 301
Treated | 298 | 299
Completed | 59 (Number Completed includes participants who completed base study and participants who entered into study extension.) | 34 (Number Completed includes participants who completed base study and participants who entered into study extension.)
Not Completed | 239 | 267
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 16 | 17
Not completed — Physician Decision | 11 | 7
Not completed — Sponsor Decision | 168 | 179
Not completed — Withdrawal by Subject | 35 | 34
Not completed — Other | 6 | 30
Period: Extension Study (Week 144 to 168)
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Started (Subset of participants who completed the base study may have been eligible to enter the study extension.) | 21 | 27
Completed | 0 | 1
Not Completed | 21 | 26
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor Decision | 20 | 25
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF | Total
Number analyzed (Participants) | 298 | 301 | 599
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.7 (11.0) | 35.7 (10.9) | 35.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 71 | 148
  Male | 221 | 230 | 451
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 123 | 112 | 235
  Not Hispanic or Latino | 171 | 184 | 355
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 16 | 20 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 86 | 90 | 176
  White | 171 | 169 | 340
  More than one race | 23 | 19 | 42
  Unknown or Not Reported | 0 | 1 | 1
Baseline Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Level [Count of Participants; unit: Participants] — The Abbott RealTime polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. Participants were stratified into the following baseline HIV-1 RNA levels: ≤100,000 copies/mL, >100,000 copies/mL or missing.
  Participants
    ≤100,000 copies/mL | 244 | 239 | 483
    >100,000 copies/mL | 54 | 60 | 114
    Missing | 0 | 2 | 2
Baseline Cluster of Differentiation 4+ (CD4+) T-Cell Count [Count of Participants; unit: Participants] — Plasma CD4+ T-cell count was measured in cells/mm^3 for baseline by a central laboratory. Baseline measurements were defined as the Day 1 value of each participant. Participants were stratified into the following baseline CD4+ T-cell counts: <200 cells/mm^3, ≥200 cells/mm^3, or missing.
  Participants
    <200 cells/mm^3 | 61 | 60 | 121
    ≥200 cells/mm^3 | 237 | 239 | 476
    Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) <50 Copies/mL at Week 48
Description: The Abbott RealTime polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 was presented using the Food and Drug Administration (FDA) Snapshot missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of study intervention. Participants were included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 88.9 | 88.3
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Non-Inferiority — Non-inferiority was concluded if the upper bound of the 2-sided multiplicity-adjusted 95% confidence interval (95%CI) was less than 10 percentage points; Treatment Difference = 0.46, 95% CI 2-sided [-4.73 to 5.60] — Estimated differences, CIs, & p-value for treatment differences in percent response were calculated using Miettinen & Nurminen method stratified by stratum with CMH weights; multiplicity-adjusted 95% CI corresponds to 1-sided Type 1 error of 0.02495

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE) up to Week 48
Description: An AE was any untoward medical occurrence in a study participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The percentage of participants who experienced at least one AE up to Week 48 was reported. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 48 weeks
Population: All randomized participants who received at least one dose of study intervention. Participants were included in the treatment group corresponding to the study intervention received. The final analysis for this outcome is presented here.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 90.6 | 86.3
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — Difference between treatment groups (Group 1: DOR/ISL and Group 2: BIC/FTC/TAF); Percentage Difference = 4.3, 95% CI 2-sided [-0.8 to 9.6] — Miettinen & Nurminen method was used to generate percentage difference and the associated 95%CI

3. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE up to Week 48
Description: An AE was any untoward medical occurrence in a study participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The percentage of participants who discontinued study treatment due to an AE up to Week 48 were reported. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 48 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 7.4 | 3.3
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — Difference between treatment groups (Group 1: DOR/ISL and Group 2: BIC/FTC/TAF); Percentage Difference = 4.0, 95% CI 2-sided [0.4 to 7.9] — Miettinen & Nurminen method was used to generate percentage difference and the associated 95%CI

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 96 was presented using the FDA Snapshot missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 51.7 | 57.9
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Non-Inferiority — Non-inferiority was concluded if the upper bound of the 2-sided multiplicity-adjusted 95% confidence interval (95%CI) was less than 10 percentage points. The multiplicity-adjusted 95% CI is shown corresponding to a 1-sided Type 1 error of 0.02495. The estimated differences, CIs and p-value for the treatment differences in percent response were calculated using the Miettinen and Nurminen method stratified by stratum with Cochran-Mantel-Haenszel (CMH) weights; p = 0.945, Miettinen and Nurminen method — The estimated differences, CIs and p-value for the treatment differences in percent response were calculated using the Miettinen and Nurminen method stratified by stratum with Cochran-Mantel-Haenszel (CMH) weights; Estimated Difference = -6.42, 95% CI 2-sided [-14.21 to 1.46] — Treatment difference for DOR/ISL group minus BIC/FTC/TAF group

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 144
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 144 was presented using the Data as Observed (DAO) missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 144
Population: All randomized participants who received at least one dose of study intervention and had data available for this outcome measure at Week 144. Participants were included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 39 | 41
Percentage of participants | 64.1 | 82.9
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — Type of statistical test 'other' denotes no hypothesis testing was conducted. The CIs for the treatment differences in percent response were calculated using the Miettinen and Nurminen method stratified by stratum with Cochran-Mantel-Haenszel (CMH) weights; Estimated Difference = -19.5, 95% CI 2-sided [-38.0 to 0.2] — Treatment difference for DOR/ISL group minus BIC/FTC/TAF group

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA <40 copies/mL was determined. The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <40 copies/mL at Week 48 was presented using the FDA Snapshot missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 88.6 | 86.3
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Non-Inferiority — Non-inferiority was concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI was less than 10 percentage points; Treatment Difference = 2.12, 95% CI 2-sided [-3.23 to 7.48] — The estimated differences, CIs and p-value for the treatment differences in percent response were calculated using the Miettinen and Nurminen method stratified by stratum with Cochran-Mantel-Haenszel (CMH) weights

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA <200 copies/mL was determined. The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 48 was presented using the FDA Snapshot missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 89.6 | 88.6
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Treatment Difference = 0.83, 95% CI 2-sided [-4.25 to 5.90] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 Copies/mL at Week 96
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <40 copies/mL at Week 96 was presented using the FDA Snapshot missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 51.0 | 57.5
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — Type of statistical test 'other' denotes no hypothesis testing was conducted. The estimated differences, and confidence intervals (CIs) for the treatment differences in percent response were calculated using the Miettinen and Nurminen method stratified by stratum with Cochran-Mantel-Haenszel (CMH) weights; Estimated Difference = -6.74, 95% CI 2-sided [-14.53 to 1.15] — Treatment difference for DOR/ISL group minus BIC/FTC/TAF group

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 96
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 96 was presented using the FDA Snapshot missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 52.3 | 58.5
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — [test comment as in outcome 8, analysis 1]; Estimated Difference = -6.41, 95% CI 2-sided [-14.20 to 1.46] — Treatment difference for DOR/ISL group minus BIC/FTC/TAF group

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 Copies/mL at Week 144
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <40 copies/mL at Week 144 was presented using the DAO missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 144
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 39 | 41
Percentage of participants | 64.1 | 82.9
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — [test comment as in outcome 5, analysis 1]; Estimated Difference = -19.5, 95% CI 2-sided [-38.0 to 0.2] — Treatment difference for DOR/ISL group minus BIC/FTC/TAF group

11. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 144
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 144 was presented using the DAO missing data approach. The final analysis for this outcome is presented here.
Time Frame: Week 144
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 39 | 41
Percentage of participants | 64.1 | 82.9
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — [test comment as in outcome 5, analysis 1]; Estimated Difference = -19.5, 95% CI 2-sided [-38.0 to 0.2] — Treatment difference for DOR/ISL group minus BIC/FTC/TAF group

12. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 4+ (CD4+) T-Cell Counts at Week 48
Description: Plasma CD4+ T-cell count was measured in cells/mm^3 for baseline and at Week 48 by a central laboratory. Baseline measurements were defined as the Day 1 value of each participant. The mean change from baseline in CD4+ T-cell count at Week 48 using the Data as Observed (DAO) approach was presented. The final analysis for this outcome is presented here.
Time Frame: Baseline (Day 1) and Week 48
Population: All randomized participants who received at least one dose of study intervention and had data available, including baseline data available for CD4+ T-cell count at Week 48. Participants were included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 263 | 263
cells/mm^3 | 182.4 [162.0 to 202.7] | 233.5 [211.8 to 255.3]

13. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 4+ (CD4+) T-Cell Counts at Week 96
Description: Plasma CD4+ T-cell count was measured in cells/mm^3 for baseline and at Week 96 by a central laboratory. Baseline measurements were defined as the Day 1 value of each participant. The mean change from baseline in CD4+ T-cell count at Week 96 using the Data as Observed (DAO) approach was presented. The final analysis for this outcome is presented here.
Time Frame: Baseline (Day 1) and Week 96
Population: All randomized participants who received at least one dose of study intervention and had data available, including baseline data available for CD4+ T-cell count at Week 96. Participants were included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 159 | 168
cells/mm^3 | 217.05 [187.52 to 246.58] | 319.92 [290.53 to 349.32]
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — Type of statistical test 'other' denotes no hypothesis testing was conducted. The CIs for mean difference in CD4+ T-cell count change from baseline were based on analysis of covariance (ANCOVA) models adjusted by baseline CD4+ T-cell count, stratum, and treatment group; Mean Difference (Final Values) = -91.75, 95% CI 2-sided [-132.59 to -50.90] — Treatment Difference (DOR/ISL minus BIC/FTC/TAF)

14. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 4+ (CD4+) T-Cell Counts at Week 144
Description: Plasma CD4+ T-cell count was measured in cells/mm^3 for baseline and at Week 144 by a central laboratory. Baseline measurements were defined as the Day 1 value of each participant. The mean change from baseline in CD4+ T-cell count at Week 144 using the Data as Observed (DAO) approach was presented. The final analysis for this outcome is presented here.
Time Frame: Baseline (Day 1) and Week 144
Population: All randomized participants who received at least one dose of study intervention and had data available, including baseline data available for CD4+ T-cell count at Week 144. Participants were included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 24 | 32
cells/mm^3 | 239.6 [177.4 to 301.8] | 350.9 [265.7 to 436.1]
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — [test comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = -111.8, 95% CI 2-sided [-218.8 to -4.8] — Treatment Difference (DOR/ISL minus BIC/FTC/TAF)

15. Secondary Outcome: Incidence of Viral Resistance-Associated Substitutions (RASs) at Week 48
Description: RASs was defined as participants with confirmed HIV-1 RNA ≥200 copies/mL and/or genotypic or phenotypic analysis of data showing evidence of resistance to the study drug administered. The number of participants who demonstrated RASs at Week 48 was presented. The final analysis for this outcome is presented here.
Time Frame: Week 48
Population: Participants with data available at Week 48. Per protocol, participants who met the definition of confirmed virologic rebound or incomplete virologic response, or who discontinued study intervention for another reason and had HIV-1 RNA ≥200 copies/mL at the time of discontinuation. Among such participants, those with HIV-1 RNA ≥400 copies/mL were included. Participants for whom available genotypic or phenotypic data showed evidence of resistance, irrespective of viral load, were also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 3 | 6
Participants | 1 | 0

16. Secondary Outcome: Incidence of Viral RASs at Week 96
Description: RASs was defined as participants with confirmed HIV-1 RNA ≥200 copies/mL and/or genotypic or phenotypic analysis of data showing evidence of resistance to the study drug administered. The number of participants who demonstrated RASs at Week 96 was presented. The final analysis for this outcome is presented here.
Time Frame: Week 96
Population: Participants with data available at Week 96. Per protocol, participants who met the definition of confirmed virologic rebound or incomplete virologic response, or who discontinued study intervention for another reason and had HIV-1 RNA ≥200 copies/mL at the time of discontinuation. Among such participants, those with HIV-1 RNA ≥400 copies/mL were included. Participants for whom available genotypic or phenotypic data showed evidence of resistance, irrespective of viral load, were also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 5 | 9
Participants | 2 | 0

17. Secondary Outcome: Incidence of Viral RASs at Week 144
Description: RASs was defined as participants with confirmed HIV-1 RNA ≥200 copies/mL and/or genotypic or phenotypic analysis of data showing evidence of resistance to the study drug administered. The number of participants who demonstrated RASs at Week 144 was presented. The final analysis for this outcome is presented here.
Time Frame: Week 144
Population: Participants with data available at Week 144. Per protocol, participants who met the definition of confirmed virologic rebound or incomplete virologic response, or who discontinued study intervention for another reason and had HIV-1 RNA ≥200 copies/mL at the time of discontinuation. Among such participants, those with HIV-1 RNA ≥400 copies/mL were included. Participants for whom available genotypic or phenotypic data showed evidence of resistance, irrespective of viral load, were also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 5 | 9
Participants | 2 | 0

18. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 48
Description: Body weight was measured at baseline and at Week 48. Participants removed their shoes and wore a single layer of clothing at each measurement. Baseline measurements were defined as the Day 1 value of each participant. The mean change from baseline in body weight at Week 48 was presented. The final analysis for this outcome is presented here.
Time Frame: Baseline (Day 1) and Week 48
Population: All randomized participants who received at least one dose of study intervention and had data available, including baseline data available, for this outcome measure at Week 48. Participants were included in the treatment group corresponding to the study intervention received. The final analysis for this outcome is presented here.
Measure: Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 270 | 268
kilogram | 3.45 [2.83 to 4.06] | 3.32 [2.68 to 3.96]
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Superiority — Superiority will be concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI was less than 0; p = 0.73, ANCOVA; A 2-sided p-value was calculated using the Analysis of covariance (ANCOVA) model; Treatment Difference = 0.15, 95% CI 2-sided [-0.71 to 1.02] — ANCOVA model was used to generate treatment difference and the associated 95%CI. The 95% CIs for treatment difference were calculated from ANCOVA models with terms for baseline weight, sex, race, stratum, and treatment

19. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 96
Description: Body weight was measured at baseline and at Week 96. Participants removed their shoes and wore a single layer of clothing at each measurement. Baseline measurements were defined as the Day 1 value of each participant. The mean change from baseline in body weight at Week 96 was presented. The final analysis for this outcome is presented here.
Time Frame: Baseline (Day 1) and Week 96
Population: All randomized participants who received at least one dose of intervention and had data available, including baseline data available, for this outcome measure at Week 96. Participants were included in the treatment group corresponding to the study intervention received. The final analysis for this outcome is presented here.
Measure: Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 189 | 201
kilogram | 3.31 [2.45 to 4.18] | 4.13 [3.15 to 5.11]
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Superiority — Superiority will be concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI was less than 0. The CIs for treatment difference were calculated from ANCOVA models with terms for baseline weight, sex, race, stratum and treatment; p = 0.268, ANCOVA; A 2-sided p-value was calculated using the Analysis of covariance (ANCOVA) model; Estimated Difference = -0.74, 97% CI 2-sided [-2.19 to 0.71] — The CIs for treatment difference were calculated from ANCOVA models with terms for baseline weight, sex, race, stratum and treatment. The CIs at week 96 is 97% corresponds to a 1-sided Type 1 error of 0.015

20. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 144
Description: Body weight was measured at baseline and at Week 144. Participants removed their shoes and wore a single layer of clothing at each measurement. Baseline measurements were defined as the Day 1 value of each participant. The mean change from baseline in body weight at Week 144 was presented. The final analysis for this outcome is presented here.
Time Frame: Baseline (Day 1) and Week 144
Population: All randomized participants who received at least one dose of study intervention and had data available, including baseline data available, for this outcome measure at Week 144. Participants were included in the treatment group corresponding to the study intervention received. The final analysis for this outcome is presented here.
Measure: Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 40 | 42
kilogram | 4.55 [2.40 to 6.70] | 3.55 [-1.46 to 8.56]
Statistical Analysis 1: Comparison: Group 1: DOR/ISL vs Group 2: BIC/FTC/TAF; Test type: Other — Type of statistical test 'other' denotes no hypothesis testing was conducted. The CIs for treatment difference were calculated from ANCOVA models with terms for baseline weight, sex, race, stratum and treatment; Estimated Difference = 1.08, 95% CI 2-sided [-4.07 to 6.24] — The CIs for treatment difference were calculated from ANCOVA models with terms for baseline weight, sex, race, stratum and treatment

21. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a study participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The percentage of participants who experienced at least one or more AEs is presented. Per protocol, pregnancy-related AEs collected for enrolled participants are reported separately and are presented in the AE module. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 47 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 96.6 | 94.0

22. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a study participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The percentage of participants who discontinued study intervention due to an AE is presented. Per protocol, pregnancy-related AEs collected for enrolled participants are reported separately and are presented in the AE module. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 38 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: DOR/ISL | Group 2: BIC/FTC/TAF
Number analyzed (Participants) | 298 | 299
Percentage of participants | 14.1 | 9.0

ADVERSE EVENTS:
Time Frame: Up to approximately 47 months
Description: All-cause mortality: all randomized participants; AEs: all randomized participants who got ≥1 dose of study drug. Both reported for base study & open-label extension. Per protocol, "post treatment follow up" denotes participants monitored after drug discontinuation with drops in CD4+/ total lymphocyte count. Per protocol, infant serious AEs (febrile convulsion & exomphalos) & pregnancy-related AEs were collected on pregnant participants enrolled; included by the arms that participants enrolled.
Groups:
- Group 1: DOR/ISL Base Study Week 0 - Week 48; Group 1: DOR/ISL Base Study Week 48-Week 96; Group 1: DOR/ISL Base Study Week 96-Week 144; Group 1: DOR/ISL Open-Label Extension Week 144-Week 168; Group 1: DOR/ISL Post-Treatment Follow-Up: Treatment-naïve participants living with human immunodeficiency virus-1 (HIV-1) that had not received ≤10 days of prior antiretroviral therapy received blinded fixed dose combination (FDC) Doravirine/Islatravir (DOR/ISL) (100 mg doravirine [DOR]/0.75 mg islatravir [ISL]) and placebo to Bictegravir/Tenofovir Alafenamide/Emtricitabine (BIC/FTC/TAF) once daily (QD) from Day 1 to Week 96, and open-label DOR/ISL up to Week 144. At Week 144, participants who consent to enter the optional open-label study extension continued to receive open-label QD FDC of DOR/ISL (100 mg/0.75 mg) for an additional 24 weeks, up to Week 168.
- Group 2: BIC/FTC/TAF Base Study Week 0 - Week 48; Group 2: BIC/FTC/TAF Base Study Week 48 - Week 96; Group 2: BIC/FTC/TAF Base Study Week 96 - Week 144; Group 2: BIC/FTC/TAF Open-Label Extension Week 144 - Week 168; Group 2: BIC/FTC/TAF Post-Treatment Follow-Up: Treatment-naïve participants living with HIV-1 that had not received ≤10 days of prior antiretroviral therapy received blinded BIC/FTC/TAF (50 mg bictegravir [BIC], 200 mg emtricitabine [FTC], 25 mg tenofovir alafenamide [TAF]) and placebo to FDC DOR/ISL QD from Day 1 to Week 96, and open-label BIC/FTC/TAF up to Week 144. At Week 144, participants who consent to enter the optional open-label study extension continued to receive QD BIC/FTC/TAF (50 mg/200 mg/25 mg) for an additional 24 weeks, up to Week 168.
Arm/Group | Group 1: DOR/ISL Base Study Week 0 - Week 48 | Group 1: DOR/ISL Base Study Week 48-Week 96 | Group 1: DOR/ISL Base Study Week 96-Week 144 | Group 2: BIC/FTC/TAF Base Study Week 0 - Week 48 | Group 2: BIC/FTC/TAF Base Study Week 48 - Week 96 | Group 2: BIC/FTC/TAF Base Study Week 96 - Week 144 | Group 1: DOR/ISL Open-Label Extension Week 144-Week 168 | Group 2: BIC/FTC/TAF Open-Label Extension Week 144 - Week 168 | Group 1: DOR/ISL Post-Treatment Follow-Up | Group 2: BIC/FTC/TAF Post-Treatment Follow-Up
All-Cause Mortality (participants affected / at risk) | 2/298 | 0/266 | 0/146 | 0/301 | 0/267 | 0/143 | 0/21 | 0/27 | 1/112 | 0/128
Serious Adverse Events (participants affected / at risk) | 19/298 | 14/266 | 3/146 | 16/299 | 13/267 | 1/143 | 0/21 | 0/27 | 3/112 | 1/128
Other Adverse Events (participants affected / at risk) | 146/298 | 115/266 | 42/146 | 141/299 | 124/267 | 37/143 | 3/21 | 2/27 | 8/112 | 2/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DOR/ISL Base Study Week 0 - Week 48 (N=298) | Group 1: DOR/ISL Base Study Week 48-Week 96 (N=266) | Group 1: DOR/ISL Base Study Week 96-Week 144 (N=146) | Group 2: BIC/FTC/TAF Base Study Week 0 - Week 48 (N=299) | Group 2: BIC/FTC/TAF Base Study Week 48 - Week 96 (N=267) | Group 2: BIC/FTC/TAF Base Study Week 96 - Week 144 (N=143) | Group 1: DOR/ISL Open-Label Extension Week 144-Week 168 (N=21) | Group 2: BIC/FTC/TAF Open-Label Extension Week 144 - Week 168 (N=27) | Group 1: DOR/ISL Post-Treatment Follow-Up (N=112) | Group 2: BIC/FTC/TAF Post-Treatment Follow-Up (N=128)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exomphalos (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphogranuloma venereum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DOR/ISL Base Study Week 0 - Week 48 (N=298) | Group 1: DOR/ISL Base Study Week 48-Week 96 (N=266) | Group 1: DOR/ISL Base Study Week 96-Week 144 (N=146) | Group 2: BIC/FTC/TAF Base Study Week 0 - Week 48 (N=299) | Group 2: BIC/FTC/TAF Base Study Week 48 - Week 96 (N=267) | Group 2: BIC/FTC/TAF Base Study Week 96 - Week 144 (N=143) | Group 1: DOR/ISL Open-Label Extension Week 144-Week 168 (N=21) | Group 2: BIC/FTC/TAF Open-Label Extension Week 144 - Week 168 (N=27) | Group 1: DOR/ISL Post-Treatment Follow-Up (N=112) | Group 2: BIC/FTC/TAF Post-Treatment Follow-Up (N=128)
Diarrhoea (Gastrointestinal disorders) | 26 (28) | 6 (7) | 2 (2) | 20 (21) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 42 (45) | 20 (21) | 2 (2) | 47 (49) | 29 (29) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 15 (16) | 14 (14) | 4 (4) | 15 (18) | 11 (11) | 4 (4) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 17 (21) | 7 (12) | 3 (3) | 16 (24) | 17 (24) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 28 (35) | 12 (13) | 1 (1) | 25 (28) | 14 (17) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 27 (28) | 64 (75) | 25 (29) | 12 (12) | 55 (62) | 24 (27) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 19 (19) | 2 (2) | 0 (0) | 18 (18) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (17) | 11 (12) | 2 (3) | 14 (16) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 31 (36) | 13 (14) | 2 (2) | 34 (38) | 13 (15) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 13 (14) | 4 (4) | 1 (1) | 19 (20) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04233879/Prot_SAP_001.pdf